CLINICAL TRIAL: NCT00110721
Title: A Phase II, Multi-Center, Open-Label Trial to Evaluate the Efficacy and Safety of Intravenous GM-CT-01 in Combination With 5-Fluorouracil When Administered in Monthly Cycles as Third- or Fourth-Line Therapy for Metastatic Colorectal Cancer
Brief Title: GM-CT-01 Plus 5-Fluorouracil as Third- or Fourth-Line Therapy for Metastatic Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study protocol amended to a new treatment regimen: study DAVFU-006.
Sponsor: Galectin Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAVFU-003
Record Dates: First submitted 2005-05-12; First posted 2005-05-13 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2012-03

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; DAVANAT; 5-fluorouracil
MeSH Terms: conditions — Colorectal Neoplasms | interventions — galactomannan; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GM-CT-01 plus 5-Fluorouracil — Single use vials, combined regimen of GM-CT-01 / 5-Fluorouracil (280 mg/m2 /500 mg/m2) given for 4 consecutive days in a 28 day cycle until disease progression.
  Other Names: DAVANAT

SUMMARY:
This is a Phase II, multi-center study of GM-CT-01 which has been shown to increase the anti-tumor activity of 5-fluorouracil (5-FU) in mice. 5-FU is a chemotherapy drug commonly used in cancer patients. In this Phase II study, patients with colon cancer which has spread, despite treatment with approved therapies, will receive GM-CT-01 plus 5-FU in monthly cycles for at least 2 cycles or until their disease progresses.

DETAILED DESCRIPTION:
A Phase I study of 40 patients showed that GM-CT-01 in different doses plus 5-FU was well tolerated in patients with different types of solid tumors who failed standard, approved treatments. The main reason for doing this Phase II study in advanced colorectal cancer patients is to verify the safety observations in the early Phase I study and further evaluate the efficacy of these drugs' combination to stabilize tumors, preventing further growth and potentially shrink tumors.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Has a histologically-proven adenocarcinoma of the colon or rectum
* Has documentation of locally advanced or metastatic colorectal cancer not amenable to curative surgery or radiotherapy
* Eligible subjects are those whose unresectable, locally advanced and/or metastatic colorectal cancer has progressed during or after receiving treatment with at least two, but not more than three, lines of therapy that collectively must have included at a minimum all of the following agents: 5-fluorouracil or capecitabine, irinotecan, and oxaliplatin (unless, in the opinion of the investigator, the subject is not able to receive irinotecan and/or oxaliplatin due to medical contraindications, in which case irinotecan and/or oxaliplatin are not required to have been included in the prior lines of therapy). Adjuvant chemotherapy following definitive management of the primary lesion in the colon or rectum is allowed and will not be counted as a line of therapy.
* Has 1 or more measurable lesion(s) ("target lesion[s]") according to RECIST (Response Evaluation Criteria in Solid Tumors) criteria.

The same diagnostic imaging method must be used throughout the study to evaluate the lesions; and clinically detected lesions will only be considered measurable when they are superficial (e.g., skin nodules and palpable lymph nodes).

* Has an ECOG performance status of 0-2
* Has a life expectancy greater than 3 months
* Has the ability to understand the nature of the study and any hazards of participating in it; to communicate satisfactorily with the Investigator; and to participate in, and comply with, the requirements of the entire study
* A female of childbearing potential must have a negative serum screening test for pregnancy and agree to practice abstinence or use an effective method of contraception
* Has had all aspects of the protocol explained and written informed consent obtained

Exclusion Criteria:

* Has central nervous system metastasis
* Has bony metastasis as the sole metastasis
* Has other concomitant or previous malignancy in the past 3 years, except:

  * adequately treated in situ carcinoma of the uterine cervix;
  * basal or squamous cell carcinoma of the skin; and/or
  * melanoma in situ.
* Is receiving concomitant anti-neoplastic treatment; has received radiation therapy in the past 3 weeks; has been treated with anti-angiogenesis agents, including bevacizumab, in the past 4 weeks; or has been treated with any other chemotherapeutic agents in the past 4 weeks (6 weeks for mitomycin C and nitrosoureas).
* Has an active infection
* Has congestive heart failure (Class III or IV in the New York Heart Association functional classification system)
* Has a hemoglobin level of < 8.5 gm/dL
* Has a platelet count of < 100,000/mm3
* Has a neutrophil count of < 1,500/mm3
* Has a serum creatinine level of > 2.0 mg/dL
* Has liver aminotransferase and alkaline phosphatase levels that are > 2.5 times the laboratory's upper limit of normal (ULN) in a subject with no liver metastases, and levels that are > 5 times the laboratory's ULN in a subject with liver metastases
* Has a total bilirubin level that is > 2 times the laboratory's ULN
* Has pulmonary DLCO < 60% of predicted
* Has known or clinically suspected infection with human immunodeficiency virus (HIV)
* Has participated within 30 days, or will participate concurrently, in another investigational drug or vaccine study
* Has a history of drug or alcohol dependence in the past 3 years
* Has other serious, non-malignant, significant, acute or chronic medical or psychiatric illness that, in the judgment of the Investigator, could compromise subject safety, limit the subject's ability to complete the study, and/or compromise the objectives of the study
* Has known intolerance to 5- FU
* Has previously participated in a GM-CT-01 clinical trial
* Has known hypersensitivity to GM-CT-01 or any of its components

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-05; Primary Completion 2007-06 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
frequency of objective complete or partial tumor response | 20 patients completed treatment
  Tumor response as characterized by Response Evaluation Criteria in Solid Tumors (RECIST) criteria
frequency of stable disease | 20 patients completed treatment
  Stable disease as measured by CT imaging or carcinoembryonic antigen (CEA) levels

SECONDARY OUTCOMES:
safety of GM-CT-01 plus 5-FU | 20 patients completed treatment
  Frequency and type of AE/SAE and ancillary clinical indicators including Eastern Cooperative Oncology Group (ECOG) performance and quality of life.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (4):
  - Medical Oncology and Hematology, Waterbury, Connecticut
  - Hematology-Oncology Associates of the Treasure Coast, Port Saint Lucie, Florida
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
- Israel (2):
  - Soroka University Medical Center, Beersheba
  - Shaare Zedek Medical Center, Oncology, Jerusalem

REFERENCES:
- See also: Sponsor's website — http://www.pro-pharmaceuticals.com